CLINICAL TRIAL: NCT00454051
Title: Double Blind Placebo Controlled Study to Assess the Expression of IgE on Basophils and Dendritic Cells During Omalizumab Treatment.
Brief Title: Effect of Omalizumab on Expression of IgE Receptors in Adults With Severe, Inadequately Controlled Allergic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIGE025AFR02
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Results first posted 2011-08-01 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Asthma, anti-immunoglobulin E, omalizumab, IgE receptors
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab (Active Comparator): Omalizumab was injected subcutaneously every 2 weeks or every 4 weeks for 16 weeks. Dose and dosing interval were determined based on patient body weight and pre-treatment serum IgE level.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Placebo was injected subcutaneously every 2 weeks or every 4 weeks for 16 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a sterile, freeze dried preparation, to be reconstituted to deliver 150mg of omalizumab. Each vial was reconstituted with 1.4ml of sterile water for injection. The appropriate dose and dosing frequency of omalizumab were determined by baseline total IgE and body weight. A dosing table was used following the European Summary of Product Characteristics (SmPC) of omalizumab.
  Arms: Omalizumab
Drug: placebo — Placebo was a physiological salt solution, administered according to the same administration scheme to respect the same dosing frequency and injected volume.
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the expression of IgE high affinity receptors (the part of the cell associated with allergic response) in patients suffering from uncontrolled severe asthma despite long term treatment with high dose of inhaled corticosteroid and long acting Beta-2 agonist.

DETAILED DESCRIPTION:
Double blind placebo controlled study to assess the expression of IgE on blood basophils and dendritic cells in patients with uncontrolled, severe, persistent allergic asthma after a 16-week Omalizumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >= 18 years.
* Patients with severe persistent allergic asthma with the following characteristics:
* FEV1 (Forced Expiratory Volume in One Second) <80% of predicted.
* Frequent daily symptoms (>=4 days/week on average) or nocturnal awakening (>=1/week on average).
* Multiple severe asthma exacerbations: either >=2 severe asthma exacerbations having required an unscheduled medical intervention with systemic corticosteroid in the past year, or hospitalization (including emergency room treatment) for an asthma exacerbation in the past year.
* Despite a high dose inhaled corticosteroid >1000 mg beclomethasone dipropionate or equivalent and a inhaled long-acting B2-agonist.
* With an allergy to a perennial allergen demonstrated with convincing criteria, i.e. positive prick skin test or in vitro reactivity to a perennial aeroallergen (RAST).
* Total serum IgE level >= 30 to <=700 IU/ml and suitable serum total IgE level and weight according to Xolair dosing tablets.

Exclusion Criteria:

* Age < 18 years.
* Smoking history > 20 pack years.
* Patients who have had an asthma exacerbation during the 4 weeks prior to randomization
* History of food or drug related severe anaphylactoid or anaphylactic reaction
* Elevated serum IgE levels for reasons other than allergy (e.g. parasite infections, hyperimmunoglobulin E syndrome, Wiskott-Aldrich Syndrome or allergic bronchopulmonary aspergillosis).
* Patients with active cancer, suspicion of cancer or any history of cancer.
* Pregnant women.
* Known hypersensitivity to omalizumab or to one of its components.
* Patients already treated with omalizumab (indeed a previous treatment with omalizumab could have modified the FceRI expression).
* Patients who had participated in a clinical trial in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigator site, Rueil-Malmaison, France

REFERENCES:
- [Derived] Chanez P, Contin-Bordes C, Garcia G, Verkindre C, Didier A, De Blay F, de Lara MT, Blanco P, Moreau JF, Robinson P, Bourdeix I, Trunet P, Le Gros V, Humbert M, Molimard M. Omalizumab-induced decrease of FcxiRI expression in patients with severe allergic asthma. Respir Med. 2010 Nov;104(11):1608-17. doi: 10.1016/j.rmed.2010.07.011. Epub 2010 Aug 30. PMID 20801010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 20 | 11
Completed | 17 | 8
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 20 | 11 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.30) | 50.6 (16.31) | 47.4 (14.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change (%) From Baseline in FcεRI (High-affinity IgE Receptor) Expression on Blood Basophils and Dendritic Cells After 16 Weeks of Treatment With Omalizumab as Compared With Placebo
Description: Blood was drawn from participants at baseline and at Week 16. Basophils and dendritic cells expressing FcεRI were counted and the percentage was calculated. Fluorescence was used to label FcεRI so that they could be visualized. The greater the fluorescence intensity the greater FcεRI expression. The change from baseline is described by the difference (%) between the baseline value, before the first study drug administration, and the value observed at the end of study, expressed as a percent of the baseline value.
Time Frame: Baseline and Week 16
Population: The Intent-to-treat (ITT) population analyzable for FcεRI expression was a subset of the ITT population and included the 27 participants with accurate measurements before and after 16 weeks of treatment.
Measure: Mean (Standard Deviation); unit: percent change in FcεRI expression
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 16 | 11
percent change in FcεRI expression
  % Change in Basophils expressing FcεRI | -0.1 (8.39) | 3.9 (7.00)
  % Change in Dendritic cells expressing FcεRI | -5.9 (27.14) | 14.8 (22.80)

2. Secondary Outcome: Change (%) From Baseline in Percent of Basophils and Dendritic Cells Expressing FcεRI After 4, 8, 12 and 16 Weeks of Treatment
Description: Blood was drawn from a sub-group of participants at weeks 4, 8, 12, and 16. Basophils and dendritic cells expressing FcεRI were counted and the percentage was calculated. Fluorescence was used to label FcεRI so that they could be visualized. The change from baseline is described by the difference (%) between the baseline value, before the first study drug administration, and the value observed at the specified time point, expressed as a percent of the baseline value.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: A subset of the ITT population analyzable for FcεRI expression at select sites had repeat measurements of FcεRI expression at all time points.
Measure: Mean (Standard Deviation); unit: percent change in cells expressing FcεRI
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 8 | 4
percent change in cells expressing FcεRI
  % change Basophils expressing FcεRI at Week 4 | 1.9 (7.89) | -5.2 (8.46)
  % change Basophils expressing FcεRI at Week 8 | 2.5 (8.60) | 0.9 (1.49)
  % change Basophils expressing FcεRI at Week 12 | 3.7 (23.49) | -6.4 (11.92)
  % change Basophils expressing FcεRI at Week 16 | 4.6 (9.40) | -1.4 (3.29)
  % change Dendritic cells expressing FcεRI Week 4 | -16.1 (33.54) | -4.7 (17.73)
  % change Dendritic cells expressing FcεRI Week 8 | -1.9 (14.66) | 6.2 (7.03)
  % change Dendritic cells expressing FcεRI Week 12 | -10.3 (19.62) | -2.8 (27.98)
  % change Dendritic cells expressing FcεRI Week 16 | -9.8 (11.07) | 23.0 (24.70)

3. Secondary Outcome: Change (%) From Baseline in the Mean Fluorescence Intensity of FcεRI After 4, 8, 12 and 16 Weeks of Treatment
Description: as for outcome 2
Time Frame: Baseline, Weeks 4, 8, 12, and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change in fluorescence intensity
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 8 | 4
% change in fluorescence intensity
  % change on basophils at Week 4 | -85.1 (6.09) | -45.8 (41.14)
  % change on basophils at Week 8 | -81.0 (9.08) | -11.5 (40.83)
  % change on basophils at Week 12 | -86.8 (6.36) | -24.2 (60.18)
  % change on basophils at Week 16 | -88.6 (4.39) | 54.2 (11.71)
  % change on dendritic cells at Week 4 | -38.6 (42.76) | -36.6 (27.95)
  % change on dendritic cells at Week 8 | -27.1 (40.13) | -12.2 (42.56)
  % change on dendritic cells at Week 12 | -31.2 (60.61) | -14.1 (55.42)
  % change on dendritic cells at Week 16 | -49.2 (30.21) | 47.1 (92.44)

4. Secondary Outcome: Change From Baseline in the Number of Days With Asthma Symptoms Per Week
Description: Participants maintained a diary to record the number of days with daytime asthma symptoms per week. This analysis compares the mean number of days per week with asthma symptoms during the 4-week screening period prior to randomization with the mean number of days per wek with asthma symptoms in the last 4 weeks of study treatment (Weeks 12 -16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: The intent-to-treat population included all randomized participants who received at least one dose of study drug and from whom at least one efficacy measurement was obtained.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
days per week
  Baseline | 5.9 (1.71) | 4.5 (2.26)
  Change from Baseline | -2.3 (2.77) | -0.9 (1.79)

5. Primary Outcome: Change (%) From Baseline in Mean Fluorescence Intensity of FcεRI After 16 Weeks of Treatment With Omalizumab as Compared With Placebo
Description: as for outcome 1
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in fluorescence intensity
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 16 | 11
percent change in fluorescence intensity
  % Change in Basophil fluorescence intensity | -77.5 (20.83) | 20.0 (76.70)
  % Change in Dendritic cell fluorescence intensity | -41.4 (36.90) | 36.7 (101.66)

6. Secondary Outcome: Change From Baseline in the Number of Puffs of Rescue Medication Per Week
Description: Participants maintained a diary to record the daytime number of puffs of rescue Short-acting B2 agonist (SABA) used to treat asthma symptoms per week. This analysis compares the mean number of puffs of rescue medication per week during the 4 week screening period prior to randomization to the mean number of puffs per week during the last 4 weeks on study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: puffs per week
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
puffs per week
  Baseline | 19.7 (24.68) | 10.5 (13.43)
  Change from Baseline | -2.0 (16.13) | -2.7 (7.75)

7. Secondary Outcome: Change From Baseline in the Number of Nights With Awakenings Per Week
Description: Participants maintained a diary to record the number of nights with awakenings due to asthma symptoms per week. For this analysis, the mean number of nights with awakenings per week during the 4 week screening period prior to randomization was compared with the mean number of nights with awakenings per week during the last 4 weeks of study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nights with awakenings per week
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
nights with awakenings per week
  Baseline | 2.5 (2.55) | 1.7 (2.15)
  Change from Baseline | -1.2 (2.08) | -0.4 (1.31)

8. Secondary Outcome: Change From Baseline in the Number of Days With Impairment in Daily Activities Per Week
Description: Impairment was defined as days with physical activity considered as limited (or "not normal") according to patient's assessment and was recorded in a patient daily diary. For this analysis, the mean number of days with impairment per week during the 4 week screening period prior to randomization was compared with the mean number of days with impairment per week during the last 4 weeks on study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
days per week
  Baseline | 4.9 (2.35) | 4.5 (2.41)
  Change from Baseline | -1.6 (2.43) | -1.0 (2.53)

9. Secondary Outcome: Change From Baseline in the Number of Days With Absence From School or Work Due to Asthma Symptoms
Description: Participants maintained a diary to record the number of days with absence from school or work due to asthma symptoms. For this analysis, the number of days with absence from school or work in the four weeks prior to randomization (screening period) were compared with the number of absence days during the last 4 weeks on study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
days
  Baseline | 2.7 (7.38) | 2.5 (8.44)
  Change from Baseline | -0.9 (2.54) | 0.1 (0.30)

10. Secondary Outcome: Change From Baseline in the Number of Days With Hospitalizations
Description: Participants maintained a diary to record the number of days with hospitalizations during the study. For this analysis, the number of days with hospitalizations during the screening period (4 weeks prior to randomization) was compared with the number of days with hospitalizations during the last 4 weeks on study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
days
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Change from Baseline | 0.0 (0.0) | 0.0 (0.0)

11. Secondary Outcome: Change From Baseline in the Number of Unscheduled Clinic Visits
Description: Participants maintained a diary to record the number of unscheduled clinic visits during the study. For this analysis, the number of unscheduled visits during the 4 week screening period prior to randomization is compared with the number of unscheduled visits during the last 4 weeks on treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: unscheduled visits
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
unscheduled visits
  Baseline | 0.2 (0.62) | 0.1 (0.30)
  Change from Baseline | -0.1 (0.55) | 0.1 (0.54)

12. Secondary Outcome: Change From Baseline in the Morning Daily Peak Expiratory Flow (PEF)
Description: Peak Expiratory Flow (PEF) was measured every morning using a peak flow meter, and was recorded in the patient diary. For this analysis, the mean morning PEF during the 4-week screening period prior to randomizaton is compared with the mean morning PEF during the last 4 weeks of study treatment (Weeks 12 - 16).
Time Frame: Baseline (the 4 week screening period prior to randomization) and End of Study (Weeks 12 - 16)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 20 | 11
liters per minute
  Baseline | 303.5 (122.07) | 317.8 (77.37)
  Change from Baseline | 9.9 (54.06) | 10.5 (28.8)

13. Secondary Outcome: Physician's Overall Assessment of Treatment Effectiveness
Description: The Physician's overall assessment of treatment effectiveness was graded 1-5 as 1 = Excellent asthma control (complete control) 2 = Good asthma control (marked improvement) 3 = Moderate asthma control (discernible, but limited improvement) 4 = Poor asthma control (no appreciable change) 5 = Very poor asthma control (worsening)
Time Frame: After 16 weeks of treatment
Population: The ITT population included all randomized participants who received at least one dose of study drug and from whom at least one efficacy measurement was obtained. Complete data for 26 of the total 30 participants was recorded.
Measure: Number; unit: participants
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 17 | 9
participants
  Excellent | 3 | 1
  Good | 5 | 2
  Moderate | 6 | 4
  Poor | 3 | 1
  Worsening | 0 | 1

ADVERSE EVENTS:
Arm/Group | Omalizumab | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/11
Other Adverse Events (participants affected / at risk) | 13/20 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=20) | Placebo (N=11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=20) | Placebo (N=11)
Conjunctivitis (Eye disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.